CLINICAL TRIAL: NCT05577130
Title: Growth Pattern and Characteristics of Cardiac Pediatric Patients Attending Assiut University Children Hospital and Sidi Galal Health Insurance Clinic
Brief Title: Growth Pattern and Characteristics of Cardiac Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Ahmed Mohamed, Resident doctor in family medicine, Assiut University
Other Study IDs: GPACOCPAAUCHASGHIC
Record Dates: First submitted 2021-09-16; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Growth Disorders
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) is the most common congenital anomaly in the body, affecting about 8 per 1000children. cardiovascular disorders are the most debilitating and one of causes of organic growth disorders in children.Malnutrition is a constant phenomenon among children with CHD. The degree and type of malnutrition may be related to characteristics of the CHD, including presence of cyanosis, congestive heart failure (CHF), or pulmonary hypertension (PHTN).

DETAILED DESCRIPTION:
At birth, the weight and length of children with CHD are close to normal and APGAR scores are generally high. Cyanotic patients are affected in growth, depending on the severity of tissue hypoxemia and on the degree of physiological variation. Mostly acute malnutrition occurs in a cyanotic heart disease but chronic malnutrition occurs in cyanotic lesions. The severity of malnutrition variety from mild under nutrition to failure to thrive. impairing growth and increasing post-operative morbidity and mortality. Early rapid growth retardation detection in early age and improved nutritional status have the potential to reduce cardiac impact on growth and feeding. Insure appropriate nutrition in those patients by the two main methods (enteral and parenteral) help in better outcome

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-4 years old
* Male and female,
* diagnosed as cardiac diseased children

Exclusion Criteria:

* children more than 4 years old
* not genetic disorder as down syndrome This is a descriptive study.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Age: 0-4 years old
  * Male and female
  * diagnosed as cardiac patient
  * children are not more than 4 years old.
  * Not genetic disorder as down syndrome
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Study the pattern of growth in infant and children with heart diseases. | through study completion, an average of 1 year.
  By measurement of :
  * Weight in (Kg)and height in (m) will be combined to report BMI in kg/m^2).
  * Measure mid arm circumference in (cm) & head circumference in(cm)

REFERENCES:
- [Background] Arodiwe I, Chinawa J, Ujunwa F, Adiele D, Ukoha M, Obidike E. Nutritional status of congenital heart disease (CHD) patients: Burden and determinant of malnutrition at university of Nigeria teaching hospital Ituku - Ozalla, Enugu. Pak J Med Sci. 2015 Sep-Oct;31(5):1140-5. doi: 10.12669/pjms.315.6837. PMID 26649002
- [Background] Mari MA, Cascudo MM, Alchieri JC. Congenital Heart Disease and Impacts on Child Development. Braz J Cardiovasc Surg. 2016 Feb;31(1):31-7. doi: 10.5935/1678-9741.20160001. PMID 27074272
- [Background] El-Koofy N, Mahmoud AM, Fattouh AM. Nutritional rehabilitation for children with congenital heart disease with left to right shunt. Turk J Pediatr. 2017;59(4):442-451. doi: 10.24953/turkjped.2017.04.011. PMID 29624225
- [Background] Venugopalan P, Akinbami FO. Anthropometric measurements in children with congenital heart disease. Trop Doct. 2001 Jul;31(3):186-8. doi: 10.1177/004947550103100333. No abstract available. PMID 11444357
- [Background] Blasquez A, Clouzeau H, Fayon M, Mouton JB, Thambo JB, Enaud R, Lamireau T. Evaluation of nutritional status and support in children with congenital heart disease. Eur J Clin Nutr. 2016 Apr;70(4):528-31. doi: 10.1038/ejcn.2015.209. Epub 2015 Dec 23. PMID 26695725
- [Background] Secker DJ, Jeejeebhoy KN. How to perform Subjective Global Nutritional assessment in children. J Acad Nutr Diet. 2012 Mar;112(3):424-431.e6. doi: 10.1016/j.jada.2011.08.039. Epub 2012 Mar 1. PMID 22717202